CLINICAL TRIAL: NCT03601728
Title: A Personalized Medicine Prehabilitation Intervention Delivered Using Wearable Mobile Devices to Improve Cognitive Function in Elective Joint Replacement Surgery
Brief Title: A Personalized Prehabilitation Intervention In Elective Joint Replacement Surgery
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 Crisis
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Carsten Skarke, MD, MD, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 826962
Record Dates: First submitted 2018-05-03; First posted 2018-07-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Arthropathy of Knee Joint; Arthropathy of Hip Joint
Keywords: elective

STUDY DESIGN:
Intervention Model Description: Matched case-control study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Monitoring Program (Experimental): Four weeks prior to the scheduled (elective) surgery, participants will receive a 60-minute in person education session how to increase the level of physical activity. This will be followed by 4 weeks of keeping this level of physical activity, which will be monitored and supported by personalized interactive prompts delivered by a smartwatch. This approach is called personalized prehabilitation.
  Interventions: Behavioral: personalized prehabilitation
- Regular Monitoring Program (No Intervention): Participants randomized to this arm will receive standard perioperative care.

INTERVENTIONS:
Behavioral: personalized prehabilitation — The 60-minute education session includes a 30-minute general education on exercise in older adults and a 30-minute instruction on participating in the study intervention (how to work with the personalized circadian-based activity guideline). The education session will be developed and presented by the PI and the certified exercise trainer. The general education session will be designed using materials from Go4Life program from the National Institute on Aging (https://go4life.nia.nig.gov). The personalized circadian-based activity guideline (exercise goal and plan) will be developed by the investigators and the exercise trainer based on the individual's typical daily circadian profile, functional status, preference for exercise.
  Other Names: Enhanced Monitoring Program
  Arms: Enhanced Monitoring Program

SUMMARY:
The mission is to develop novel interventions to improve cognitive function, and thereby reducing delirium in hospitalized patients to improve perioperative outcomes. Delirium affects up to 42% of hospitalized patients and disproportionately increases morbidity and mortality in older adults, especially after surgical procedures. Current approaches prevent only 30-40% of delirium cases. The goal is to use prehabilitation (an individualized exercise regimen performed in the 2-4 weeks prior to admission) to improve peri-operative cognitive status, mobility and recovery. Based on preliminary data, the investigators propose to deeply phenotype patients, meaning to study the patient, the disease and surgery in a very detailed fashion, with elective knee or hip replacement surgery and use a personalized prehabilitation intervention compared to standard pre-operative care. To facilitate data collection over the course of the study, the investigators use wearable devices and mobile phone applications.

DETAILED DESCRIPTION:
The fiscal burden estimated at $164 billion annually in the US alone, with delirium often leading to significant increases in hospital length of stay. The pathophysiology of delirium is multifactorial and incompletely understood. Disruption of circadian rhythms, with subsequent impairment of alertness, and increased inflammation including neuroinflammation, is common in hospital environments, and is associated with poorer outcome, particularly in the elderly.

An intriguing new therapeutic concept currently emerging in the area of elective surgery is prehabilitation, a form of exercise training, which when pre-emptively administered in the weeks prior to admission, has the potential to improve postoperative cognitive status, mobility and recovery, thereby minimizing complications such as delirium. Our team has recently developed a novel personalized medicine intervention that uses wearable devices (smartwatches) to create an individualized exercise regimen for older adults that can facilitate prehabilitation and monitor adherence to the prehabilitation regimen while the patient is at home. In one sense, prehabilitation can be conceptualized as bouts of physical exercise performed at home prior to admission, which, when adequately timed using guidance by a wrist-worn biometric mobile device (smartwatch), augment the robustness of circadian rhythms, particularly in the elderly. This intervention has the potential to have a high impact because of its low cost, personalized nature, and ability to monitor adherence to confirm maximization of functional status prior to admission.

ELIGIBILITY:
Inclusion Criteria:

* Adults scheduled for elective arthroplasty;
* ≥55 years of age;
* Capable of giving informed consent;
* Willing to comply either to undergo prehabilitation (cases) or standard preoperative care (control);
* Own a smartphone.

Exclusion Criteria:

* Patients with bilateral or revision surgeries;
* Diagnosis of pre-existing dementia;
* Test result of <20 in the MoCA indicating moderate to severe dementia;
* Diagnosis of acute stroke;
* Diagnosis of neurologic injury;
* Current alcohol (more than 2 drinks a day with last drink within the past 3 days) or substance abuse (positive urine dip test for illicit drugs) history at risk of postoperative withdrawal;
* Active diagnosis of alcohol or substance abuse;
* Recent travel across more than two (2) time zones (within the past month);
* Planned travel across more than two (2) time zones during the planned study activities;
* Subjects, who have received an experimental drug, used an experimental medical device within 30 days prior to screening, or who gave a blood donation of ≥ one pint within 8 weeks prior to screening;
* Subjects without access to WiFi in their or close to home or at work.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline, pre-prehabilitation cognitive function at 30±2 days post-operative | 30±2 days post-operative
  Difference in cognitive function as assessed by the CogState Brief Battery for the condition 'baseline, pre-prehabilitation' versus 30±2 days post-operative between Intervention vs. Control

SECONDARY OUTCOMES:
Change from baseline, pre-prehabilitation physical activity [vector magnitude] at 30±2 days post-operative | 30±2 days post-operative
  Difference in physical activity for the condition 'baseline, pre-prehabilitation' versus 30±2 days post-operative between Intervention vs. Control
Change from baseline, pre-prehabilitation step count [number] at 30±2 days post-operative | 30±2 days post-operative
  Difference in step count for the condition 'baseline, pre-prehabilitation' versus 30±2 days post-operative between Intervention vs. Control
Change from baseline, pre-prehabilitation sleep duration [hours] at 30±2 days post-operative Difference in sleep parameters | 30±2 days post-operative
  Difference in sleep duration for the condition 'baseline, pre-prehabilitation' versus 30±2 days post-operative between Intervention vs. Control
Change from baseline, pre-prehabilitation circadian phase [hours] of activity | 30±2 days post-operative
  Difference in circadian phase for the condition 'baseline, pre-prehabilitation' versus 30±2 days post-operative between Intervention vs. Control
Change from baseline, pre-prehabilitation circadian amplitude [difference between the maximum and minimum observed values] of activity | 30±2 days post-operative
  Difference in circadian phase for the condition 'baseline, pre-prehabilitation' versus 30±2 days post-operative between Intervention vs. Control
Compliance | 2 months
  Compliance to the four-week prehabilitation paradigm assessed as the delta between the first and fourth (last) week of physical activity in the intervention group
Difference in incidence of delirium | 30±2 days post-operative
  Difference in incidence of delirium between Intervention vs. Control assessed from patient charts at 'post-operative day 30±2'
Difference in concentrations of Interleukin-6 (IL-6) [pg/mL] | 30±2 days post-operative
  Difference in concentrations between Intervention vs. Control
Difference in concentrations of S100β [ng/mL] | 30±2 days post-operative
  Difference in concentrations between Intervention vs. Control
Difference in hospital length of stay | 30±2 days post-operative
  Difference in hospital length of stay [days] for Intervention vs. Control

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Skarke, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
to be determined

REFERENCES:
- [Background] Skarke C, Lahens NF, Rhoades SD, Campbell A, Bittinger K, Bailey A, Hoffmann C, Olson RS, Chen L, Yang G, Price TS, Moore JH, Bushman FD, Greene CS, Grant GR, Weljie AM, FitzGerald GA. A Pilot Characterization of the Human Chronobiome. Sci Rep. 2017 Dec 7;7(1):17141. doi: 10.1038/s41598-017-17362-6. PMID 29215023
- See also: Study support by the Penn Center for Precision Medicine (PCPM) — https://lp.pennmedicine.org/precision-medicine/general?hcmacid=pm
- See also: Study description in a 1-minute YouTube video — https://www.youtube.com/watch?v=XpEu03PQM0Q